CLINICAL TRIAL: NCT06323980
Title: Randomized, Prospective, Multi-Center Study of the INHANCE Stemless Total Reverse Shoulder System
Brief Title: INHANCE Stemless Reverse Shoulder IDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSM202108; DSM202108 (Other: DePuy Orthopaedics)
Record Dates: First submitted 2024-02-27; First posted 2024-03-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Arthroplasty; Replacement; Shoulder
Keywords: Reverse Shoulder; Stemless Shoulder; Total Shoulder

STUDY DESIGN:
Intervention Model Description: 2:1 Randomized (Stemless to Stemmed)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- INHANCE Stemless Reverse (Experimental): INHANCE(TM) Stemless Reverse Total Shoulder
  Interventions: Device: Reverse Total Shoulder
- INHANCE Stemmed Reverse (Active Comparator): INHANCE(TM) Stemmed Reverse Total Shoulder
  Interventions: Device: Reverse Total Shoulder

INTERVENTIONS:
Device: Reverse Total Shoulder — Uncemented Reverse Total Shoulder

SUMMARY:
2:1 Randomized, Controlled, Multi-Center, Prospective, Pre-Market Study of the INHANCE Stemless Reverse Cementless Total Shoulder.

DETAILED DESCRIPTION:
There is one primary effectiveness endpoint and there are three primary safety endpoints:

1. Primary effectiveness endpoint - Adjusted Constant-Murley Change from Baseline (ACM CFB) at 2 years post-operative
2. Primary safety endpoint(s):

   1. No revision, removal, reoperation, supplemental fixation, or other intervention for any system component
   2. No humeral or glenoid radiolucent line >2 mm is present in 50% or more zones at 2 years
   3. No conclusive evidence of migration and tilt (>5mm migration and >10° tilt) of the humeral or glenoid component at 2 years

The study will be successful if the primary effectiveness endpoint non-inferiority analysis is successfully demonstrated, and no significant difference is seen on any of the 3 primary safety endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals requiring reverse total shoulder replacement for a severely painful, disabling, arthritic joint (i.e. osteoarthritis, post-traumatic arthritis and rotator cuff arthropathy).
2. Individuals who are anatomically and structurally suited to receive the implants and have a functional deltoid muscle.
3. Individuals who are able to read and comprehend the informed patient consent document and are willing and able to provide informed patient consent for participation in the study and have authorized the transfer of their information to DePuy Synthes.
4. Individuals who are willing and able to return for follow-up as specified by the study protocol.
5. Individuals who are a minimum age of 22 years at the time of consent.
6. Individuals who are willing and able to complete the Patient Reported Outcome Measure questionnaires (PROMs) as specified by the study protocol.

Exclusion Criteria:

1. BMI > 40 kg/m2
2. Individuals have active, uncontrolled local infection or systemic infection.
3. Patients who have not reached skeletal maturity, regardless of age.
4. Either preoperatively or intraoperatively and per standard of care medical assessment, bone stock in the proximal humerus or glenoid fossa is determined to be inadequate for supporting the INHANCE humeral stemless components (NOTE: exclusion applies to both arms of the study, i.e., bone stock to be evaluated independent of randomized treatment assignment).
5. Intraoperatively and per treating physician's assessment of bone quality, bone is determined to be too soft or porous to support the implant or that is too hard or brittle to allow for proper bone preparation and fixation, i.e. osteoporosis or sclerotic bone, or tumor(s) of the supporting bone structure, where there could be considerable migration of the prosthesis and/or a chance of fracture of the humerus or glenoid.
6. Fractures of the proximal humerus that could compromise the fixation of the INHANCE reverse humeral stemless components.
7. Patients who have undergone previous treatment on the study shoulder that may compromise fixation of the INHANCE reverse humeral stemless component.
8. Revision of a failed hemi, total or reverse shoulder arthroplasty.
9. Patient is receiving, or is scheduled to receive, treatment that the Investigator considers could affect bone quality, such as chemotherapy or high dose corticosteroids.
10. Individuals who are bedridden per the Investigator's determination.
11. Individuals that have participated in a clinical investigation with an investigational product (drug or device) in the last three months.
12. Individuals currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
13. Individuals, in the opinion of the Investigator, who are drug or alcohol abusers or have psychological disorders that could affect their ability to complete patient reported questionnaires or be compliant with follow-up requirements.
14. Patients with a known medical condition that the Investigator believes would impact the study outcomes (including, but not limited to osteomyelitis, Paget's disease, neuropathies such as Charcot's disease, metastatic or neoplastic disorders).
15. Patient has a medical condition with less than 2 years life expectancy.
16. Patients who are known to be pregnant or breastfeeding.
17. Known polyethylene and/or metal sensitivity or allergy.
18. Contralateral side has been enrolled in the study or has received a total shoulder operation within the last 6 months
19. Otherwise determined by the investigator to be medically unsuitable for participation in this study
20. Patient is a member of a vulnerable population (i.e., incarcerated individuals - those incarcerated for at least one month and considered to be an inmate)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2027-11-10 (Estimated); Study Completion 2028-09-29 (Estimated)

PRIMARY OUTCOMES:
Constant Murley Score (CMS) | Pre-op, 2 years
  Primary effectiveness endpoint - Adjusted Constant-Murley Change from Baseline (ACM CFB) at 2 years post-operative. The CMS is a 100 point scale, the higher the score, the higher the quality of the function. ACM will be obtained by dividing the raw score by the relative score.
Removal of any system component | 2 year
  No removal of any system component
Revision of any system component | 2 year
  No revision of any system component
Reoperation of any system component | 2 year
  No reoperation of any system component
Supplemental Fixation of any system component | 2 year
  No supplemental fixation of any system component
Radiolucent Lines (Humeral & Glenoid) | 2 year
  No humeral or glenoid radiolucent line greater than 2mm is present in 50% or more zones
Migration and Tilt (Humeral & Glenoid) | 2 year
  No conclusive evidence of migration and tilt (greater than 5mm migration and greater than 10 degrees tilt) of the humeral or glenoid component

SECONDARY OUTCOMES:
Constant Murley Score (CMS) | Pre-op, 3-month, 6-month, 1 year, 2 year
  Adjusted Constant-Murley Score at baseline and 3- and 6-months and 1- and 2-years post-operative. The CMS is a 100 point scale, the higher the score, the higher the quality of the function. ACM will be obtained by dividing the raw score by the relative score.
EQ-5D-5L and EQ-VAS | Pre-op, 3-month, 6-month, 1 year, 2 year
  EQ-5D-5L Scores by dimension and EQ-VAS, at baseline and 3- and 6-months and 1- and 2-years post-operative. The value score generally ranges from less than 0 to 1, with higher scores indicating higher health utility. The EQ VAS records the subject's self-rated health from 0 (worst) to 100 (best).
Simple Shoulder Test | Pre-op, 3-month, 6-month, 1 year, 2 year
  Simple Shoulder Test (SST) Scores at baseline and 3- and 6-months and 1- and 2-years post-operative. Scores range from 0 (worst) to 12 (best).
Single Assessment Numeric Evaluation (SANE) Score | Pre-op, 3-month, 6-month, 1 year, 2 year
  Single Assessment Numeric Evaluation (SANE) Scores at baseline and 3- and 6-months and 1- and 2-years post-operative. The scale is 0 to 100 with 100 being "normal".
Survivorship | 2 year
  Overall survivorship of the INHANCE Shoulder System at 2 years post-operative, where the system is deemed to be surviving if no components (humeral stem or stemless component, glenosphere, baseplate, liner, etc.) have been removed for any reason, will be presented using the Kaplan-Meier method.
Complications | 2 year
  The type and frequency of all reportable adverse events (AEs) and device deficiencies in this study will be summarized, with distinction of serious AEs, device and procedure related AEs

OTHER OUTCOMES:
Constant Murley Score (CMS) | Pre-op, 3-month, 6-month, 1 year
  Change from baseline adjusted Constant-Murley Score at 3- and 6-months and 1- year post-operative. The CMS is a 100 point scale, the higher the score, the higher the quality of the function. ACM will be obtained by dividing the raw score by the relative score.
EQ-5D-5L and EQ-VAS | Pre-op, 3-month, 6-month, 1 year, 2 year
  Change from baseline EQ-5D-5L Value Score and EQ-VAS, at 3- and 6-months and 1- and 2-years post-operative. The value score generally ranges from less than 0 to 1, with higher scores indicating higher health utility. The EQ VAS records the subject's self-rated health from 0 (worst) to 100 (best).
Simple Shoulder Test | Pre-op, 3-month, 6-month, 1 year, 2 year
  Change from baseline SST Scores at 3- and 6-months and 1- and 2-years post-operative. Scores range from 0 (worst) to 12 (best).
Single Assessment Numeric Evaluation (SANE) Score | Pre-op, 3-month, 6-month, 1 year, 2 year
  Change from baseline SANE Scores at 3- and 6-months and 1- and 2-years post-operative. The scale is 0 to 100 with 100 being "normal".
Range of Motion | Pre-op, 3-month, 6-month, 1 year, 2 year
  Change from baseline range of motion at 3- and 6-months and 1- and 2-years post-operative

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Hoag Orthopedic Institute, Irvine, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Orthopedic Center of Palm Beach County, Atlantis, Florida
  - Boston Sports & Shoulder Center, Waltham, Massachusetts
  - Trinity Health Grand Rapids, Grand Rapids, Michigan
  - Missouri Orthopaedic Institute (MOI), Columbia, Missouri
  - OrthoCarolina Research Institute Charlotte, Charlotte, North Carolina
  - Duke Orthopaedics of Raleigh, Raleigh, North Carolina
  - Crystal Clinic Orthopaedic Center, Akron, Ohio
  - Lindner Research Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Slocum Center for Orthopaedics and Sports Medicine, Eugene, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Rothman Orthopaedics Institute, Philadelphia, Pennsylvania
  - MTBJ a division of Tennessee Orthaepedic Alliance, Columbia, Tennessee
  - TOSH- The Orthopedic Specialty Hospital, Murray, Utah
  - University of Utah, Salt Lake City, Utah